CLINICAL TRIAL: NCT04412525
Title: Comparative Study 27G Vitrectomy vs Larger Gauge Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S63610
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: Vitreoretinal Surgery
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 27 gauge needle vitrectomy surgery (Active Comparator): ultra-small gauge
  Interventions: Device: vitrectomy (27G gauge or larger needle)
- larger than 27 gauge (23G or 25G) needle vitrectomy surgery (Active Comparator): 23-gauge and 25-gauge instruments are a little larger in size
  Interventions: Device: vitrectomy (27G gauge or larger needle)

INTERVENTIONS:
Device: vitrectomy (27G gauge or larger needle) — vitrectomy surgery for either floater removal or macular surgery, with or without combined cataract (phaco) surgery.
  Other Names: vitrectomy surgery with 27G or larger needle technique

SUMMARY:
Two-arm, mono-center, prospective, interventional comparative case study to compare postoperative recovery between the 27G and larger gauge surgical approach.

DETAILED DESCRIPTION:
A prospective randomized comparison of postoperative recovery between 27-gauge and larger gauge surgical approaches to evaluate efficiencies and postoperative outcomes of the surgical gauges. Fifty patients who were scheduled to undergo pars plana vitrectomy (PPV) for floaters or macular surgery were treated with either 27-gauge or 23-gauge techniques and assessed for efficiency of the procedures as well as a variety of postop indicators of pain and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18
* No prior vitrectomy surgery in the study eye (for the same eye)
* No prior inclusion in this trial
* Scheduled for vitrectomy for floater removal or macular surgery (including macular holes) without endotamponades such as PFCL, Gas, Silicone oil). (Air tamponade is allowed )

Exclusion Criteria:

* • Patients with serious heart, lung, liver, or kidney dysfunction

  * Patients with proliferative diabetic retinopathy, endophthalmitis, uveitis, eyes with refraction >+5D or exceeding -8D , or other eye disease that impacts the outcome of vitrectomy surgery
  * Patients with HIV
  * Patients with history of drug abuse or alcoholism
  * Patients participating in other drug or medical device clinical trials before screening for this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-01-23 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
changes in post-operative outcome of pain | day 1 postoperative
  by assessing the amount of pain on a visual analogue scale (score 0-9)
changes in post-operative outcome of redness | day 1 postoperative
  scoring the amount of redness on a scale 0-4 through eye photos
changes in post-operative outcome in grading of anterior chamber cells | day 1 postoperative
  clinical assessment by slit lamp examination (Tyndall 0-3 and Cells 0-3)

SECONDARY OUTCOMES:
visual acuity | day 1 postoperative
  best corrected visual acuity in LogMar will be obtained to report the visual acuity
intra-ocular pressure | day 1 postoperative
  Millimeter of Mercury pressure (mmHg) will be measured to report the intra-ocular pressure
pain-assessment | 1 week postoperative
  a questionnaire with visual analogue scale will be used to assess the level of pain up to 1 week after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, PhD, Principal Investigator — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04412525/Prot_SAP_000.pdf